CLINICAL TRIAL: NCT03094884
Title: Pulsed Low Dose Rate Radiation With Concurrent Chemotherapy for Non-Small Cell Lung Cancer and Esophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-101
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer; Esophageal Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms | interventions — Heart Rate; Radiation; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pulsed Low dose radiation with Carboplatin/Paclitaxel (Experimental): Pulsed Low Dose Radiation concurrent with Carboplatin and Paclitaxel
  Interventions: Radiation: Pulsed Low Dose Radiation; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Pulsed Low Dose Radiation — Treatment naïve patients with non-small cell lung cancer or esophageal cancer whose planned treatment regimen is concurrent CRT followed by surgery. The total radiation dose will be 50.4 Gy in daily fraction of 1.8 Gy for esophageal cancer and 60 Gy in daily fraction of 2 Gy for non-small cell lung cancer. The concurrent chemo regimen will carboplatin-paclitaxel managed by the treating medical oncologist. Patients are planned to receive surgery at approximately 6 to 9 weeks after finishing CRT with surgical aspects determined by the treating surgical oncologist.
Drug: Carboplatin — Treatment naïve patients with non-small cell lung cancer or esophageal cancer whose planned treatment regimen is concurrent CRT followed by surgery. The total radiation dose will be 50.4 Gy in daily fraction of 1.8 Gy for esophageal cancer and 60 Gy in daily fraction of 2 Gy for non-small cell lung cancer. The concurrent chemo regimen will carboplatin-paclitaxel managed by the treating medical oncologist. Patients are planned to receive surgery at approximately 6 to 9 weeks after finishing CRT with surgical aspects determined by the treating surgical oncologist.
Drug: Paclitaxel — Treatment naïve patients with non-small cell lung cancer or esophageal cancer whose planned treatment regimen is concurrent CRT followed by surgery. The total radiation dose will be 50.4 Gy in daily fraction of 1.8 Gy for esophageal cancer and 60 Gy in daily fraction of 2 Gy for non-small cell lung cancer. The concurrent chemo regimen will carboplatin-paclitaxel managed by the treating medical oncologist. Patients are planned to receive surgery at approximately 6 to 9 weeks after finishing CRT with surgical aspects determined by the treating surgical oncologist.

SUMMARY:
Phase I study with the hypothesis that Pulsed Low Dose Radiation (PLDR) radiation delivery technique can significantly decrease the rate of severe acute esophagitis in patients receiving concurrent Chemo-radiation therapy (CRT) for non-small cell lung cancer or esophageal cancer while maintaining similar efficacy. For these patients, the rate of severe acute esophagitis during concurrent CRT is high (approximately 20%) when conventional external beam radiation is utilized. Severe acute esophagitis can cause many adverse consequences such as severe discomfort, weight loss, hospitalization, interruption/early termination of treatment, and worse surgical complications for those who receive surgery after CRT. PLDR radiation has the potential to maintain the tumor control rates of conventional radiation while decreasing the toxicity to the surrounding normal tissue 29-35.

We have completed accrual to a phase I PLDR radiation study, in which patient received palliative re-irradiation with PLDR technique for their metastatic disease in previous irradiated field. In that phase I study, PLDR demonstrated safety for acute toxicities in the setting of re-irradiation for a total dose of 50 Gy, with analysis of 60 Gy pending. The follow up time for that phase I study is limited as most enrolled patients have short overall survival due to their terminal illness.

This proposed phase I study is, to our knowledge, the first clinical study with combination of PLDR radiation and concurrent chemotherapy for definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have pathologically-confirmed and previously untreated:

   * Non-small cell lung cancer, Stage IIIA (T1-3 N2 M0); OR
   * Localized esophageal cancer, ≥T2, or N+, and M0 according to the American Joint Committee on Cancer (AJCC) 7th edition staging.
2. The planned treatment regimen must be concurrent chemoradiation with Carboplatin-Paclitaxel followed by surgery.
3. Age > 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status is 0-1.
5. Laboratory studies must meet each of the following criteria (with labs drawn within 4 weeks prior to the registration):

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   * Platelets ≥100,000 cells/mm3
   * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable)
   * Creatinine ≤2 X the upper limit of normal
   * Bilirubin ≤ 1.5 X upper limit of normal
   * Aspartate transaminase (AST) ≤ 3 X upper limit of normal
6. Men and women of childbearing potential must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy completed.
7. Patients must be able to read and write English to comply with the questionnaire portions of the protocol.
8. Subjects must sign a written informed study consent and HIPAA consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.

Exclusion Criteria:

1. Patients who have had previous radiotherapy in the thorax.
2. Patients who have a history of ataxia telangiectasia or other documented history of radiation hypersensitivity.
3. Patients who have a history scleroderma or other active connective tissue disease.
4. Women of childbearing potential must not be pregnant with a negative urine pregnancy test within 72 hours prior to registration and non-lactating; postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential; woman status post oophorectomy or hysterectomy are considered non-childbearing potential
5. Patients who have uncontrolled inter-current illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of severe acute esophagitis in patients with lung cancer and esophageal cancer treated with concurrent CRT using PLDR technique. | 2 years
  The investigator will evaluate the severity of other adverse events using the NCI Common Terminology Criteria for Adverse Events (CTCAE v.4.0).

SECONDARY OUTCOMES:
Quality of life | 1 year
  Quality of life will be evaluated based on a quality of life survey conducted at different time-points during the study. After entering in the study survey will be conducted in 1st month , 2nd month ,3rd month, 6th month, 9th month. Number of surveys conducted will be the same however a delay due toxicity is possible and therefore last survey could be collected up to 12 months.
Progression free survival | 1-5 years
  progression free survival will be evaluated from the day of first treatment until disease progression
Response rate based | 1 year
  Response rate will be evaluated based on the outcome of surgical pathology

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No